CLINICAL TRIAL: NCT03761368
Title: Remote Ischemic Preconditioning and Contrast Induced - Acute Kidney Injury in Patients Undergoing Elective Percutaneous Coronary Intervention - Randomised Clinical Trial
Brief Title: Remote Ischemic Preconditioning and Contrast Induced - Acute Kidney Injury in Patients Undergoing Elective PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Karolina Stokfisz, Principal Investigator, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RNN/219/13/KE
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Results first posted 2020-10-30 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2018-11

CONDITIONS: Remote Ischemic Preconditioning; Contrast Induced - Acute Kidney Injury
Keywords: remote ischemic preconditioning; contrast induced-acute kidney injury; neutrophil gelatinase-associated lipocalin; percutaneous coronary intervention

STUDY DESIGN:
Intervention Model Description: After admission to the Department, patients were randomly assigned in 1:1 ratio to either control group or RIPC - group by means of a computerized randomization table.
Who Masked: Investigator
Masking Description: Blinded investigator, not involved in either CA or randomization procedure, performed assignment intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC group (Experimental): The RIPC group underwent Remote Ischemic Preconditioning.
  Interventions: Procedure: Remote Ischemic Preconditioning
- Control group (Sham Comparator): Patients from control group had sham Remote Ischemic Preconditioning.
  Interventions: Procedure: Sham Remote Ischemic Preconditioning

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — four cycles of 5-min inflation to 200 mmHg followed by 5-min deflation of left upper - arm cuff
  Other Names: RIPC
  Arms: RIPC group
Procedure: Sham Remote Ischemic Preconditioning — deflated cuff placed on the left arm for 40 min
  Other Names: Sham RIPC
  Arms: Control group

SUMMARY:
Prospective, randomized, sham-controlled clinical study was conducted to assess whether RIPC reduces the incidence of CI-AKI measured standard way of using SCr concentration but also with the use of serum NGAL as a new potential biomarker of kidney injury. Furthermore, the aim of investigation was to analyse the safety and clinical outcomes of RIPC after elective coronary angiography (CA) followed by percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Nowadays CI-AKI is defined according to serum creatinine concentration (SCr) as any of the following: (1) an absolute rise of ≥ 0.5 mg/dL (44 µmol/L) and/or (2) a relative increase of 25% in serum creatinine compared to baseline within 48 to 72 hours after contrast administration. In the last decades, several novel biomarkers of AKI have been studied including neutrophil gelatinase-associated lipocalin (NGAL). Furthermore, remote ischemic preconditioning (RIPC) turned out to be one of the most promising and intriguing non-pharmacological strategy. This simple procedure consisting of brief, non-lethal episodes of ischemia and reperfusion applied in one tissue or organ protects remote tissues or organs from subsequent injury.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* patients with stable angina pectoris
* patients admitted to Intensive Cardiac Therapy Clinic Medical University of Lodz with intention of elective CA with follow-up PCI.

Exclusion Criteria:

* history of severe injuries up to 2 months before intervention
* history of surgeries up to 2 months before intervention
* history of cancer,
* acute inflammation during hospitalization
* chronic autoimmunologic diseases
* patients needing hemodialysis
* chronic kidney disease in stage 4 or 5 (eGFR<30 ml/min/1,73m2)
* peripheral vascular disease affecting upper limbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marzenna Zielinska, MD PhD, Study Chair — Medical University of Lodz
Locations (1):
- Intensive Cardiac Therapy Clinic, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Yes
The data sets used and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years after the end of the study
Access Criteria: on reasonable request

REFERENCES:
- [Derived] Stokfisz K, Ledakowicz-Polak A, Kidawa M, Zielinska M. Remote Ischemic Preconditioning and Contrast-Induced Acute Kidney Injury in Patients Undergoing Elective Percutaneous Coronary Intervention: A Randomized Clinical Trial. Curr Ther Res Clin Exp. 2020 Aug 5;93:100599. doi: 10.1016/j.curtheres.2020.100599. eCollection 2020. PMID 32874376

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients aged over 18 years presented with stable angina pectoris, admitted to Intensive Cardiac Therapy Clinic Medical University of Lodz and scheduled for elective CA with follow-up PCI.
Period: Overall Study
Arm/Group | RIPC Group | Control Group
Started | 50 | 51
Completed | 50 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- RIPC Group: The RIPC group underwent Remote Ischemic Preconditioning.
  Remote Ischemic Preconditioning: four cycles of 5-min inflation to 200 mmHg followed by 5-min deflation of left arm cuff
- Total: Total of all reporting groups
Arm/Group | RIPC Group | Control Group | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 23 | 25 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 33 | 33 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 51 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Contrast Medium Intake [Median (Inter-Quartile Range); unit: ml] | 100 [80 to 140] | 110 [90 to 140] | 110 [80 to 140]
Serum creatinine on admission [Median (Inter-Quartile Range); unit: µmol/L] | 87 [81 to 96] | 88 [82 to 101] | 88 [81 to 99]
NGAL on admission [Median (Inter-Quartile Range); unit: ng/mL] | 71.3 [55.8 to 86.8] | 80.6 [55.8 to 101.2] | 74.4 [55.8 to 102.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Contrast Induced-Acute Kidney Injury
Description: absolute rise of ≥ 0.5 mg/dL (44 µmol/L) and/or a relative increase of 25% in serum creatinine compared to baseline
Time Frame: 48 to 72 hours after contrast exposure
Measure: Number; unit: participants
Arm/Group | RIPC Group | Control Group
Number analyzed (Participants) | 50 | 51
participants | 2 | 3

2. Secondary Outcome: Number of Participants With Need of Renal Replacement Therapy
Description: qualification for RRT according to standard clinical criteria (level of serum creatinine, serum urea concentration, electrolytes levels (sodium, potassium, chlorides), hydration management)
Time Frame: up to 7 days after contrast exposure
Measure: Number; unit: participants
Arm/Group | RIPC Group | Control Group
Number analyzed (Participants) | 50 | 51
participants | 0 | 0

3. Secondary Outcome: Number of Participants Who Presented Cardiogenic Shock
Description: sustained hypotension (systolic blood pressure < 90 mm Hg for ≥30 min)
Time Frame: up to 7 days after contrast exposure
Measure: Number; unit: participants
Arm/Group | RIPC Group | Control Group
Number analyzed (Participants) | 50 | 51
participants | 1 | 1

4. Secondary Outcome: Death of Any Cause
Description: Number of patients who died.
Time Frame: up to one month after contrast exposure
Measure: Number; unit: participants
Arm/Group | RIPC Group | Control Group
Number analyzed (Participants) | 50 | 51
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to one month
Groups:
- RIPC Group: The RIPC group underwent Remote Ischemic Preconditioning.
  Remote Ischemic Preconditioning: four cycles of 5-min inflation to 200 mmHg followed by 5-min deflation of left upper-arm cuff
Arm/Group | RIPC Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/50 | 1/51
Other Adverse Events (participants affected / at risk) | 1/50 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RIPC Group (N=50) | Control Group (N=51)
Cardiogenic shock (Cardiac disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIPC Group (N=50) | Control Group (N=51)
skin petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — petechiae on the skin of preconditioned arm distally to upper - arm cuff placement

LIMITATIONS AND CAVEATS:
1. Single-center trial.
2. Relatively small sample size.
3. We were unable to observe sufficient number of events, such as CI-AKI, mortality, need for dialysis as an endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT03761368/SAP_001.pdf
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT03761368/Prot_002.pdf